## **PROTOCOL**

| Study Title: | Apremilast 30 mg BID combined with<br>Dupilumab for the Treatment of Recalcitrant<br>Moderate-to-Severe Atopic Dermatitis |
|---|---|
| Study Drug: | Oral Apremilast 30 mg BID |
| Sponsor: | David Rosmarin, MD Tufts Medical Center Department of Dermatology 800 Washington Street, Box 114 Boston, MA 02111 Phone: (617) 636-7462 Fax: (617) 636-9169 E-mail: drosmarin@tuftsmedicalcenter.org |
| NCT: | NCT04306965 |
| <u>Version and Date</u> : | Version June 2, 2021 |

## **Statistical Methods**

Sample size: We will screen up to 20 patients to ensure that 16 patients complete the study.

**General statistical Methods:** A clinical response to apremilast for the purposes of this study will be defined as an Investigator Global Assessment score of 0 (clear) or 1 (almost clear). The end points of the study will be assessed at Week 16. A period of 16 weeks was chosen, as this was the time frame utilized for primary endpoint reporting in the ESTEEM clinical program.<sup>6,8</sup> An additional 8 weeks of study drug will be provided to assess enhanced clinical benefit with continued use at 24 weeks. A rate of incompletion and/or drop out of subjects has been factored in to assure great than 16 patients will complete the study.

The analysis will be primarily descriptive. Mean, standard deviation, median, minimum, maximum, and 95% confidence interval for mean will be provided for continuous variables. Changes and percent changes from pre-treatment to on-treatment time points will be calculated for continuous efficacy points. Graphical displays of changes over time may be presented for key outcomes. Counts, percentages, and 95% confidence intervals will be provided for categorical variables. Subgroup analyses, such as gender stratification and stratification based on baseline treatment regimens, will be performed to identify a patient population that achieves the most benefit.

Efficacy analyses will only use data from participants who complete at least 16 weeks of study treatment in order to evaluate the primary endpoint.